CLINICAL TRIAL: NCT04536922
Title: Single Patient Protocol: A Study Using the Administration of Autologous T-Cells Genetically Engineered to Express T-Cell Receptors Reactive Against Mutated or Viral Neoantigens in a Patient With Metastatic Cancer Plus the Administration of Pembrolizumab
Brief Title: Administration of Autologous T-Cells Genetically Engineered to Express T-Cell Receptors Reactive Against Mutated or Viral Neoantigens in a Patient With Metastatic Cancer Plus the Administration of Pembrolizumab
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Subject no longer able to participate in this single pt study.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000163; 000163-C
Record Dates: First submitted 2020-09-02; First posted 2020-09-03 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Metastatic HPV-16 Positive Squamous Cell Anal Cancer
Keywords: Gene Therapy; Immunotherapy; Cell Therapy; Adoptive Cell Therapy
MeSH Terms: interventions — Cyclophosphamide; fludarabine; aldesleukin; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- iTCR + Pembro (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + Individual Patient TCR-Transduced PBL + high- or low-dose aldesleukin + pembrolizumab prior to cell administration and 3 additional doses every 3 weeks following cell infusion
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin; Drug: Pembrolizumab (KEYTRUDA(R)); Biological: Individual Patient TCR-Transduced PBL

INTERVENTIONS:
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day x 2 days IV in 250 mL D5W infused simultaneously with mesna 15 mg/kg /day over 1 hour x 2 days.
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg /m2/day IVPB daily over 30 minutes for 5 days.
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 10 doses).
Drug: Pembrolizumab (KEYTRUDA(R)) — Pembrolizumab 2 mg /kg IV over approximately 30 minutes on Days -2, 21, 42, and 63.
Biological: Individual Patient TCR-Transduced PBL — Day 0: Cells will be infused at a dose not to exceed 1.5e11 in 400 mL intravenously on the Patient Care Unit over 20-30 minutes (2-4 days after the last dose of fludarabine).

SUMMARY:
Background:

A cancer treatment has been developed called "gene transfer" or "gene therapy." It involves taking white blood cells from a person (called apheresis), genetically modifying the cells in a lab to recognize cancer, and then giving the cells back to the person. Researchers want to see if this treatment can help people with metastatic squamous cell anal cancer.

Objective:

To see if treating cancer with a person s own white blood cells that have been genetically modified can cause tumors to shrink.

Eligibility:

People who have metastatic squamous cell anal cancer for which standard treatments have not worked.

Design:

Participants will have had a tumor biopsy and apheresis to collect white blood cells under a separate protocol.

Participants will stay at the hospital for 3 to 4 weeks. They will have an intravenous (IV) catheter placed in a large vein in the upper chest.

Participants will get chemotherapy drugs (fludarabine and cyclophosphamide), the cell infusion, and aldesleukin through the IV. Pembrolizumab is given before and for three doses given every three weeks after the cell infusion. Aldesleukin will help the cells grow.

Participants will take an antibiotic, antiviral, and antifungal by mouth. They will get an injection of filgrastim. It will stimulate the formation of white blood cells.

Participants will have blood and urine tests. They will have physical exams. Their symptoms will be reviewed. They will have imaging scans.

About 6 and 12 weeks after they finish treatment, participants will have safety follow-up visits. These visits will take 1 to 2 days.

Participants will return to the Clinical Center every 3 to 6 months for 3 years, and then as determined by their doctor. They will be followed long term for up to 15 years on a separate study.

DETAILED DESCRIPTION:
Background:

* The administration of autologous tumor-infiltrating lymphocytes (TIL) can mediate complete, durable regressions in 20-25% of patients with metastatic melanoma. Recent studies have shown that these TIL predominantly recognize unique mutated or viral neoantigens expressed by the cancer not shared by other melanomas.
* Administration of bulk autologous TIL to patients with a variety of other solid cancers, including cancers of the gastrointestinal tract and genitourinary tract, have little if any therapeutic impact.
* Recent studies in the National Cancer Institute Surgery Branch (NCI-SB) have shown that TIL from non-melanoma solid cancers can also contain T-cells reactive against nonshared unique mutated neoantigens expressed in the cancer. The frequency of these Tcells is very low (often < 0.1%) and it is thus difficult to isolate and grow mutation reactive T-cells to levels required for effective therapy.
* In a single patient with chemo-refractory metastatic cholangiocarcinoma, we were able to grow a relatively pure population of neoantigen reactive TIL and administration of these cells mediated a near-complete regression of all metastatic disease now lasting 2.5 years.
* We have developed approaches to identify rare neoantigen reactive T-cells from common non-melanoma cancers, to isolate their T-cell receptors (TCR), and to genetically engineer autologous peripheral blood lymphocytes (PBL) to express these TCRs with high efficiency. The neoantigen TCR gene-modified cells can recognize and destroy the autologous cancer in vitro.
* In addition to reactivity to neoantigens derived from nonsynonymous mutations, T-cells can recognize human papilloma virus (HPV) epitopes in patients with HPV-induced cancers. The TCR from these reactive cells can be isolated and retrovirally-transduced into autologous PBL with high efficiency. This clinical protocol will treat a single patient with refractory anal cancer using the adoptive transfer of autologous PBL transduced with genes encoding TCRs that recognize unique mutated or viral neoantigens expressed by the cancer.

Objective:

-Under a single-patient IND, to treat a patient with metastatic HPV-16 positive squamous cell anal cancer with autologous peripheral blood lymphocytes (PBL) that have been transduced with genes encoding T-cell receptors that recognize mutated or viral neoantigens in the autologous cancer.

Eligibility:

* Must have measurable, metastatic disease as assessed per RECIST v1.1 criteria.
* Must sign the informed consent document.
* Willing to sign Durable Power of Attorney Form.
* Must have all regulatory approvals prior to start of treatment.

Design:

* This patient will have already undergone resection or biopsy to obtain tumor for generation of autologous TIL cultures. This will have been conducted under the NCI-SB cell harvest protocol 03-C-0277 (Cell Harvest and Preparation for Surgery Branch Adoptive Cell Therapy Protocols).
* Exomic sequencing and RNA-Seq will be performed to identify the mutations expressed in the patient s cancer. Multiple autologous TIL cultures will be grown and tested for reactivity against mutations from the autologous tumor using assays we have developed that involve the exposure of autologous antigen-presenting cells to long peptides containing the mutation or tandem mini-genes encoding the mutation.
* T-cell cultures with reactivity against mutated and viral neoantigens will be identified and the individual T-cell receptors that recognize the neoantigens will be synthesized and used to create retroviral supernatants for transduction of the TCR into the patient s autologous PBL.
* The patient will be treated with a non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine, followed by the infusion of autologous transduced PBL and then high-dose aldesleukin. The patient will also receive pembrolizumab on Day -2 prior to cell administration and three additional doses every three weeks following the cell infusion.
* Clinical and immunologic response will be evaluated about 4-6 weeks after cell infusion and periodically thereafter.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Measurable (per RECIST v1.1 criteria), metastatic squamous cell anal cancer.
2. Refractory to approved standard systemic therapy.
3. Clinical performance status of ECOG 0 or 1
4. Willing to practice birth control from the time of enrollment on this study and for four months after treatment.
5. Must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
6. Serology

   * Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive may have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
   * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
7. Hematology

   * ANC > 1000/mm^3 without the support of filgrastim
   * WBC >= 3000/mm^3
   * Platelet count >= 100,000/mm^3
   * Hemoglobin > 8.0 g/dL. Subject may be transfused to reach this cut-off.
8. Chemistry

   * Serum ALT/AST <= 5.0 x ULN
   * Serum creatinine <= 1.6 mg/dL
   * Total bilirubin <= 2.0 mg/dL, except in patients with Gilbert's Syndrome, who must have a total bilirubin < 3.0 mg/dL.
9. More than four weeks must have elapsed since completion of any prior systemic therapy at the time of enrollment. Note: Patient may have undergone minor surgical procedures or limited field radiotherapy within the four weeks prior to enrollment, as long as related major organ toxicities have recovered to grade 1 or less.
10. Ability of subject to understand and the willingness to sign a written informed consent document.
11. Willing to sign a Durable Power of Attorney Form.
12. Subject must be co-enrolled on protocol 03-C-0277.

EXCLUSION CRITERIA:

1. Patient is pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. Concurrent systemic steroid therapy.
3. Active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active or uncompensated major medical illnesses.
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and AIDS).
5. History of major organ autoimmune disease.
6. Grade 3 or 4 major organ irAEs following treatment with anti-PD-1/PD-L1, including but not limited to myocarditis and pneumonitis.
7. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immunecompetence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
8. History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or aldesleukin.
9. History of coronary revascularization or ischemic symptoms.
10. Patient is known to have an LVEF <= 45%.
11. Patient is receiving any other investigational agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Treatment | 6 and 12 weeks after cell infusion, then every 3 months x3, then every 6 months x 2 years, then per PI discretion
  Under a single-patient IND, to treat a patient with metastatic HPV-16 positive squamous cell anal cancer with autologous peripheral blood lymphocytes (PBL) that have been transduced with genes encoding T-cell receptors that recognize mutated or viral neoantigens in the autologous cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000163-C.html